CLINICAL TRIAL: NCT02455375
Title: Puumala Hantavirus Infection in France: Evaluation of Commercial Assays for the Detection of Antibodies Against This Virus and the Use of Urine Samples for the Molecular Detection of This Infection
Brief Title: Diagnostic of Puumala Virus Infection in France
Acronym: HANTADIAG
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Charleville-Mézières (Other)
Collaborators: Institut Pasteur (Industry)
Responsible Party: Sponsor
Other Study IDs: PHRC-14-0063
Record Dates: First submitted 2015-04-21; First posted 2015-05-27 (Estimated); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Nephropathia Epidemica; Hemorrhagic Fever With Renal Syndrome
Keywords: Puumala virus; diagnostic; France
MeSH Terms: conditions — Hemorrhagic Fever with Renal Syndrome; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine Plasma Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases: Case group = group of patients positive with reference tests including serological (ELISA, IF neutralization) and/or molecular assays:
  * detection of PUUV RNA in plasma collected at admission.
  * or/and detection of IgM and IgG against PUUV in serum collected at admission,
  * or/and detection of a seroconversion in IgG against PUUV from admission and late sera
- Controls: Control group = group of patients who do not have the criteria listed above

SUMMARY:
Routine Puumala virus (PUUV) infection diagnosis is performed using serological commercial kits of which performances have not been established in real life, which use recombinant protein from strains from Central or North Europe. Molecular diagnostic of these infection is not the rule. Consequently the objectives of the project are to evaluate the performances of the serological commercial assays in real life in France and to assess the use of urine versus plasma for the molecular diagnostic of this infection.

DETAILED DESCRIPTION:
Hantaviruses constitute one of the 5 genera in the family Bunyaviridae and are associated with several natural host species including rodents, insectivores and bats. Infection of these species remains unapparent. Transmission of the virus between individuals occurs through direct contact or through inhalation of saliva, feces, or urine. Using these routes, some rodent-borne hantaviruses can be transmitted to humans and cause hemorrhagic fever with renal syndrome or cardiopulmonary syndrome. Human-to-human transmission is rare. There is no specific treatment. Inactivated vaccines against Hantaan and Seoul (SEOV) viruses are only available and licensed in China and South Korea.

Puumala (PUUV), SEOV, Tula and Nova hantaviruses are reported in metropolitan France but only the 2 first are of medical importance. One single human SEOV infection has been confirmed and very few cases have been suspected. In contrast, about 100 PUUV human cases are detected yearly and occurred in the North East quarter of France.

Routine PUUV infection diagnosis is performed using serological commercial kits, allowing detection of IgM or IgG against PUUV or other hantaviruses. The performances (sensitivity and specificity) of these tests as reported by the manufacturers are very good. However, 1/ they have been established with panels of reference sera and not in real life for all assays but one; 2/ these assays are based on N recombinant protein but it has been reported that using whole virus antigens, instead of the single N protein, detection of IgG against hantavirus would be earlier; 3/ PUUV strains used to produce the recombinant N proteins are phylogenetically far from the strains detected in France, and the use of a Belgian strain close to the French strains (instead of a Scandinavian strain) since 1990 has improved the performances of the Institut Pasteur, Hantavirus National Reference Center, home-made assays.

Molecular diagnosis is not performed routinely and only 3 very recent studies reported data on PUUV viremia, using blood, plasma or sera. Urine samples previously showed to be a good alternative for PUUV detection but the use if this type of sample has not been evaluated in real life and the viruria not studied.

The performances of most of the commercial immunoassays for the detection of antibodies against hantaviruses, especially PUUV, has not yet been reported when used in real life.

The investigators propose to perform this evaluation for 9 assays, some of them now being used for the last few years by 13 French clinical laboratories:

* Euroimmun AG : Hantavirus Pool 1 " Eurasia " IgM and IgG ELISA
* Focus Diagnostics Hantavirus DxSelect IgM and IgG ELISA
* Progen Hantavirus (Puumala) IgM and IgG ELISA
* Reagena Puumala IgM and IgG EIA
* Reagena Reascan Puumala IgM (rapid test)

Furthermore, they will explore the use of urine as a sample type for molecular diagnostics. Hantaviruses are excreted in the urine of rodents and have been detected in a few studies in the urine of patients, as well as IgG and IgM against hantaviruses. The shedding of the virus may be higher and/or longer in the urine than in plasma. Viruria compared to viremia has never been reported.

The results of the study will allow the recommendation of some commercial assays to be used at admission of patients for the serological diagnosis of PUUV infection.

Furthermore, the results of the study, assessing the use of the urine versus blood for the molecular detection of PUUV, may recommend the use of the molecular techniques for the diagnostic of this infection.

ELIGIBILITY:
Inclusion Criteria:

Hospitalized patients, male or female, more than 18 years old and less than 76 years old1:

* having at admission or within 8 days preceding admission a pain , a documented febrile syndrome (body temperature ≥ 38°C) and a platelet count < 150 G/L,
* exposed to PUUV infection (for the last 6 weeks) or living in a French municipality where Hantavirus infection cases have been recorded during the 2003-2013 period or in a municipality bordering one of them ,
* giving their written consent after being informed of the research and the collection of data, and blood & urine samples.

NB: persons in emergency situation will be proposed to participate because their situation may affect the performances of laboratory diagnostics.

Exclusion Criteria:

Hospitalized patients:

* who are known to have been previously diagnosed infected by an hantavirus (medical records and/or laboratory results),
* who are known to present stable thrombocytopenia,
* who, according to the medical staff, would not adhere to the protocol,
* for whom the health status, according to the medical staff, may interfere with the study or is not compatible with the sampling planned in the study.

NB: Pregnant, parturient or breast-feeding women as well as patients under psychiatric care or patients subject to a legal protection order will be not proposed to participate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for suspected PUUV infection
Sampling Method: Non-Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients positive for the detection of IgG or IgM againt PUUV by commercial assays and by molecular/serological techniques | 33 months
  Proportion of patients tested positive for the detection of IgG or IgM against PUUV by the use of the commercial assays (index tests) and by the Hantavirus National Reference Center (NRC) molecular and serological techniques (reference tests) according to the information given in the notices of the commercial kits in use and in the version of the standard operating procedure of the Hantavirus NRC in use.

SECONDARY OUTCOMES:
Proportion of urine samples tested positive for the detection of PUUV | 33 months
  Proportion of urine samples tested positive for IgG or IgM against PUUV compare to plasma sample positive for IgG or IgM against PUUV

CONTACTS AND LOCATIONS:
Overall Officials: Jean Marc Galempoix, MD, Principal Investigator — CH de Charleville-Mézières
Locations (10):
- France (10):
  - CH Belfort-Montbéliard, Belfort
  - CHU Besançon, Besançon
  - CH Charleville Mézières, Charleville-Mézières
  - CHP Sud de l'Oise, Creil
  - CHU Dijon, Dijon
  - CH de Laon, Laon
  - CHU Reims, Reims
  - CH de Saint Claude, Saint-Claude
  - CHU Nancy, Vandœuvre-lès-Nancy
  - CH de Verdun, Verdun

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Plyusnin A, Horling J, Kanerva M, Mustonen J, Cheng Y, Partanen J, Vapalahti O, Kukkonen SK, Niemimaa J, Henttonen H, Niklasson B, Lundkvist A, Vaheri A. Puumala hantavirus genome in patients with nephropathia epidemica: correlation of PCR positivity with HLA haplotype and link to viral sequences in local rodents. J Clin Microbiol. 1997 May;35(5):1090-6. doi: 10.1128/jcm.35.5.1090-1096.1997. PMID 9114386
- [Background] Prince HE, Lieberman JM. Impact of the Yosemite hantavirus outbreak on hantavirus antibody testing at a national reference laboratory. Clin Vaccine Immunol. 2013 Aug;20(8):1213-6. doi: 10.1128/CVI.00326-13. Epub 2013 Jun 5. PMID 23740929
- [Background] Lederer S, Lattwein E, Hanke M, Sonnenberg K, Stoecker W, Lundkvist A, Vaheri A, Vapalahti O, Chan PK, Feldmann H, Dick D, Schmidt-Chanasit J, Padula P, Vial PA, Panculescu-Gatej R, Ceianu C, Heyman P, Avsic-Zupanc T, Niedrig M. Indirect immunofluorescence assay for the simultaneous detection of antibodies against clinically important old and new world hantaviruses. PLoS Negl Trop Dis. 2013 Apr 4;7(4):e2157. doi: 10.1371/journal.pntd.0002157. Print 2013. PMID 23593524
- [Background] Hentzien M, Mestrallet S, Halin P, Pannet LA, Lebrun D, Drame M, Bani-Sadr F, Galempoix JM, Strady C, Reynes JM, Penalba C, Servettaz A. Bioclinical Test to Predict Nephropathia Epidemica Severity at Hospital Admission. Emerg Infect Dis. 2018 Jun;24(6):1045-1054. doi: 10.3201/eid2406.172160. PMID 29774835
- [Result] Reynes JM, Schaeffer L, Papadopoulos P, Ait-Ahmed M, Siby-Diakite D, Ripaux-Lefevre M, Buivan TP, Lechat S, Vray M, Galempoix JM; HANTADIAG Study Group. Molecular Detection of Orthohantavirus puumalaense in Plasma and Urine Samples from Hospitalized Patients Presenting with a Serologically Confirmed Acute Hantavirus Infection in France. J Clin Microbiol. 2023 Aug 23;61(8):e0037223. doi: 10.1128/jcm.00372-23. Epub 2023 Jul 24. PMID 37486218